CLINICAL TRIAL: NCT03766386
Title: The Natural History of Danon Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Principal Investigator, Eric Adler, MD, Professor of Medicine, University of California, San Diego
Other Study IDs: 170727
Record Dates: First submitted 2018-11-30; First posted 2018-12-06 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Danon Disease
MeSH Terms: conditions — Glycogen Storage Disease Type IIb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Danon Disease Patients: Patients with a confirmed diagnosis of Danon disease who are currently alive (including patients who may or may not have undergone heart transplantation).
- Deceased Danon Disease Patients: Patients with a confirmed diagnosis of Danon disease who are deceased (including patients who may or may not have undergone heart transplantation).

SUMMARY:
Danon disease (DD) is a rare, X-linked disorder associated with severe cardiomyopathy, and in many cases, skeletal myopathy, and cognitive impairment caused by mutations in the LAMP2 gene. There is still uncertainty regarding the natural history of DD because of its rarity.

This study aims to determine the natural history of DD through the collection and analysis of retrospective and prospective data. To achieve this, the investigators will perform surveys and obtain medical records from DD patients. The same cohort of patients will also be assessed by a multidisciplinary team with expertise in DD (cardiologist, neurologist, ophthalmologist, psychologist, geneticist) at the University of California, San Diego. All patients with DD are eligible, including those who underwent a heart transplant. Additionally, data and records from deceased patients will provide valuable retrospective data for this study.

DETAILED DESCRIPTION:
The study design will include:

1. Collection of information for all patients from:

   * Survey of patient or caregiver (if the patient has deceased)
   * Medical Charts
2. Collection of information from living patients assessed by the multidisciplinary team at the University of California, San Diego including:

   * A complete medical history and physical examination
   * Cardiac Testing (Electrocardiography; Echocardiography; Cardiac magnetic resonance imaging with gadolinium contrast agent-gadolinium contrast is optional-; Cardiopulmonary Test)
   * Pulmonary function testing (PFT)
   * Neuromuscular Assessment
   * Cognitive Tests
   * Vision exam including retinal evaluation
   * Laboratory Tests
   * Questionnaires on Quality of life
   * Needle Skeletal muscle biopsy (only for patients over 18 years old)
   * Abdominal Ultrasound for assessment of the liver structure

ELIGIBILITY:
Inclusion Criteria:

• Living or deceased patients with a diagnosis of Danon disease(including patients who may or may not have undergone heart transplantation) based on a genetic test positive for the LAMP2 mutation

Exclusion Criteria:

• Patients without a genetic test positive for a LAMP2 mutation

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Danon Disease (LAMP2 mutation) of any sex and any age.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Cardiac structure over time | 6, 12, 18, 24, 30, 36 months
  Change of cardiac structure (wall thickness -mm) measured by cardiac ultrasound / cardiac magnetic resonance

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong KN, Eshraghian E, Khedro T, Argiro A, Attias J, Storm G, Tsotras M, Bloks T, Jackson I, Ahmad E, Graw S, Mestroni L, Bui QM, Schwartz J, Turner S, Adler ED, Taylor M. An International Longitudinal Natural History Study of Patients With Danon Disease: Unique Cardiac Trajectories Identified Based on Sex and Heart Failure Outcomes. J Am Heart Assoc. 2025 Apr;14(7):e038394. doi: 10.1161/JAHA.124.038394. Epub 2025 Mar 21. PMID 40118805